CLINICAL TRIAL: NCT00915577
Title: An Open-Label, Multicenter Study to Determine Subject Satisfaction in Using the Single-Use Autoinjector With a Pre-Filled Liquid AVONEX® Syringe in Multiple Sclerosis Subjects
Brief Title: Patient Satisfaction Study of Single-Use Autoinjector for the Delivery of Pre-Filled Avonex Syringe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Model: Crossover | Masking: None
Other Study IDs: C-872
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; interferon beta-1a; Avonex; liquid Avonex
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1st Injection (Experimental): Manual injection with pre-filled syringe.
  Interventions: Drug: Interferon beta-1a
- Single-use autoinjector (Experimental): Single-use autoinjector with Avonex pre-filled syringe
  Interventions: Device: Single-use autoinjector

INTERVENTIONS:
Drug: Interferon beta-1a — 30mcg, IM once-a-week
  Other Names: Avonex
  Arms: 1st Injection
Device: Single-use autoinjector — Single-use autoinjector with Avonex 30mcg pre-filled syringe
  Arms: Single-use autoinjector

SUMMARY:
Determine patient satisfaction with the single-use autoinjector for the delivery of pre-filled Avonex syringe.

ELIGIBILITY:
Inclusion Criteria:

* Must be using liquid AVONEX® to treat MS. In addition, the subject must be on liquid AVONEX® for 12 weeks prior to the Screening Visit.
* Must have a BMI of 19 to 28 kg/m², inclusive, and a minimum body weight of 50 kg at Screening.
* Must be able to physically demonstrate use of the device and be able to self-administer all injections.
* Must be English speaking.
* Must be able to understand and comply with the protocol.

Exclusion Criteria:

* Abnormal screening or screening blood tests determined to be clinically significant by the investigator for: white blood count (WBC) or differential, platelet count, hemoglobin, serum creatinine, bilirubin, alanine transaminase (ALT) aspartate transaminase (AST), prothrombin time (PT).
* Known sensitivity to dry natural rubber.
* Treatment with other agents to treat MS symptoms or underlying disease as specified in the protocol.
* History of severe allergic or anaphylactic reactions.
* History of intolerance to acetaminophen (paracetamol), ibuprofen, naproxen, and aspirin that would preclude the use of at least one of these during the study.
* Serious local infection

Other inclusion and exclusion criteria apply as per Biogen Idec Protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to determine patient satisfaction with the single-use autoinjector for the delivery of pre-filled AVONEX® syringe | The study duration is 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Study Director — Biogen